CLINICAL TRIAL: NCT01946256
Title: Erythromycin Versus Amoxicillin for Treatment of Antenatal Chlamydia Trachomatis Infection: A Randomized Controlled Trial
Brief Title: Treatment of Antenatal Chlamydia Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Obafemi Awolowo University Teaching Hospital (Other)
Responsible Party: Principal Investigator, Okunola Temitope Omoladun, Erythromycin versus Amoxicillin for treatment of antenatal Chlamydia infection: a randomized controlled trial, Obafemi Awolowo University Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC/2013/09/06
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Chlamydia Trachomatis Infection in Pregnancy
MeSH Terms: interventions — Amoxicillin; Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin (Active Comparator): Amoxicillin 500mg three times in a day for 1 week
  Interventions: Drug: Amoxicillin
- Erythromycin (Placebo Comparator): Erythromycin 500mg four times in a day for 1 week
  Interventions: Drug: Erythromycin

INTERVENTIONS:
Drug: Amoxicillin
  Arms: Amoxicillin
Drug: Erythromycin
  Arms: Erythromycin

SUMMARY:
PREGNANT WOMEN IN ANTENATAL CLINIC WILL BE SCREENED FOR CHLAMYDIA TRACHOMATIS INFECTION WITH ENDOCERVICAL SWAB.THOSE THAT TEST POSITIVE AND SATISFY THE INCLUSION CRITERIA WILL BE COUNSELLED AND ENROLLED INTO THE STUDY AFTER OBTAINING INFORMED CONSENT.THE PARTICIPANTS WILL BE RANDOMISED INTO ONE OF THE TWO GROUPS.THE DRUGS WILL BE TAKEN FOR I WEEK AND THE SEXUAL PARTNER(S) WILL ALSO BE TREATED WITH DOXYCYCLINE FOR 1 WEEK. BARRIER CONTRACEPTION WILL ALSO BE USED DURING THE TREATMENT.THE SEXUAL PARTNERS WILL BE CONTACTED THROUGH TELEPHONE CALLS AND THE BENEFITS OF PARTICIPATING IN THE STUDY WILL BE EXPLAINED TO THEM. LATEX MALE CONDOM WILL BE GIVEN TO THE WOMEN. ALSO, FOLLOW-UP TELEPHONE CALLS WILL BE PUT ACROSS TO THEM DURING THE TREATMENT WEEK TO ENHANCE COMPLIANCE. A REPEAT ENDOCERVICAL SWAB WILL BE TAKEN 4 WEEKS AFTER TREATMENT TO CHECK FOR MICROBIOLOGICAL CLEARANCE. A STUDY PROFORMA WILL BE FILLED DURING THIS VISIT. THE DATA WILL BE ANALYSED USING STATISTICAL PACKAGE FOR SOCIAL SCIENCES VERSION 17.

DETAILED DESCRIPTION:
AIM(S) OF THE RESEARCH TO ASSESS THE EFFICACY AND TOLERABILITY OF AMOXICILLIN COMPARED TO ERYTHROMYCIN IN TREATMENT OF ANTENATAL CHLAMYDIA INFECTION

OBJECTIVES OF THE RESEARCH

* TO DETERMINE THE PREVALENCE OF CHLAMYDIA TRACHOMATIS INFECTION IN PREGNANCY
* TO COMPARE THE PROPORTION OF SUBJECTS WITH CLEARANCE OF ANTENATAL CHLAMYDIA TRACHOMATIS INFECTION BETWEEN THE ERYTHROMYCIN AND AMOXICILLIN GROUPS
* TO COMPARE THE OCCURENCE OF SIDE EFFECTS BETWEEN THE TWO GROUPS
* TO COMPARE THE DRUG DISCONTINUATION RATES BETWEEN THE TWO GROUP

ELIGIBILITY:
Inclusion Criteria:

1. Test positive to Chlamydia rapid screening kit
2. Estimated gestational age less than 36 weeks
3. Consent to participate in the study
4. Willingness or ability to comply with follow-up schedule

Exclusion Criteria:

1. Antenatal patients whose gestational age is more than 36 weeks
2. History of reaction to any of the drugs
3. Women with low lying placenta or placenta Praevia
4. History of other antibiotics intake within two weeks of recruitment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
completion of course of medication and microbiological clearance | 4 weeks after treatment
  The women will be screened 4 weeks after treatment to check for microbiological clearance

SECONDARY OUTCOMES:
drug discontinuation rates | within 1 week of treatment
  The drug discontinuation rates between the two groups will be compared

OTHER OUTCOMES:
occurrence of side effect. | 1 week
  Occurrence of side effects will be considered between the two groups. The side effects include nausea, diarrhoea,vomiting and loss of appetite

CONTACTS AND LOCATIONS:
Overall Officials: Temitope O Okunola, MB;BS, Principal Investigator — Obafemi Awolowo University Teaching Hospitals Complex, Ile-Ife
Locations (1):
- Obafemi Awolowo University Teaching Hospitals Complex, Ile Ife, Ile-Ife, Imesi Ile, Nigeria

REFERENCES:
- [Background] Alary M, Joly JR, Moutquin JM, Mondor M, Boucher M, Fortier A, Pinault JJ, Paris G, Carrier S, Chamberland H, et al. Randomised comparison of amoxycillin and erythromycin in treatment of genital chlamydial infection in pregnancy. Lancet. 1994 Nov 26;344(8935):1461-5. doi: 10.1016/s0140-6736(94)90288-7. PMID 7968119